CLINICAL TRIAL: NCT06245031
Title: Open-Label Extension to a Randomized, Double-blind, Sham-controlled, Adaptive-Design Pivotal Study of Sensory Stimulation in Subjects With Alzheimer's Disease (OLE Hope Study, CA-0015)
Brief Title: Extension to a Pivotal Study of Sensory Stimulation in Alzheimer's Disease (OLE Hope Study, CA-0015)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cognito Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-0015
Record Dates: First submitted 2024-01-26; First posted 2024-02-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Cognitive Impairment; Mild Cognitive Impairment; Dementia, Mild; Dementia Moderate; Dementia Alzheimers; Dementia of Alzheimer Type; AD
Keywords: Gamma Stimulation; Cognito
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This is an Open-Label Extension of a previous randomized, sham-controlled study. All subjects in this study will receive treatment with a device with Active treatment settings. Analysis is planned to compare Active-Active treatment group to Sham-Active treatment group (delayed start model).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active (Experimental): All subjects will receive a device with Active settings for use daily at home for 60-minutes for 12 months.
  Interventions: Device: Sensory Stimulation System (GS120) - Active

INTERVENTIONS:
Device: Sensory Stimulation System (GS120) - Active — Sensory Stimulation System (GS120) - Active settings

SUMMARY:
This is an open-label extension for a multicenter, randomized, double-blind, sham-controlled, adaptive design pivotal study.

Participants who complete the Hope Study (CA-0011) will be eligible to consent for screening to enroll in the OLE Hope Study (CA-0015). All participants will be treated with an Active Sensory Stimulation System (GS120) for 60 minutes daily for up to 12 months. There will be no Sham treatment group or randomization involved in this study.

DETAILED DESCRIPTION:
This is an open-label extension for a multicenter, randomized, double-blind, sham-controlled, adaptive design pivotal study. Participants who complete the Hope Study (CA-0011) will be eligible to consent for screening to enroll in the OLE Hope Study (CA-0015). All participants will be treated with an Active Sensory Stimulation System (GS120) for 60 minutes daily for up to 12 months. There will be no Sham treatment group or randomization involved in this study.

Up to approximately 402 participants will complete the Hope Study and be offered participation in the OLE Hope Study at up to approximately 70 clinical sites.

The objective of the study will be to assess efficacy of gamma sensory stimulation (visual and audio) in slowing disease progression in the Active-Active group versus Active-Sham group for subjects with mild to moderate AD as measured functionally by the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) assessment and a combined statistical test (CST) for ADCS-ADL and the Mini-Mental State Exam (MMSE).

Participants will be treated with the Sensory Stimulation System (GS120) for 60 minutes daily for up to 12 months with Active device settings. Each participant will be involved in the study for up to 13 months: approximately 12 months of treatment and 1 month of safety follow-up.The visits in the study include: a Screening/Enrollment visit (Day 0), followed by telephone training on device receipt, a clinic visit at 12 months and a telephone visit at 6 and 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Randomized and completed 12-months of participation in the Hope Study (CA-0011)
* Non-childbearing potential or using adequate birth control
* Available/consenting Study Partner

Exclusion Criteria:

* Insufficient adherence to treatment in the Hope Study (CA-0011)
* Living in continuous care nursing home (assisted living permitted)
* Initiating or ongoing treatment with any of the following during study participation:

  * Immunomodulators or passive immunotherapies for AD (ie, monoclonal antibodies)
  * Memantine (Namenda or Namzaric)
  * Nootropic drugs except stable acetylcholinesterase inhibitors

For more information about the Hope Study (CA-0011) that participants in this study complete first, please see: https://www.hopestudyforad.com/

or the Hope Study ClinicalTrials.gov posting here: https://clinicaltrials.gov/study/NCT05637801

Ages: 50 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Function as measured by the ADCS-ADL (total score possible from 0-78, where a lower score is more affected by Alzheimer's disease)
Change from Baseline in a Combined Statistical Test (CST) that creates a composite measure (combining Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) and Mini-Mental State Exam (MMSE) scales into one measure) at 12-Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Function and Cognition as measured by CST of ADCS-ADL and MMSE (ADCS-ADL total score possible from 0-78, where a lower score is more affected by Alzheimer's disease) (MMSE total score possible from 0-30, where a lower score is more affected by Alzheimer's disease)

SECONDARY OUTCOMES:
Key Secondary: Change from Baseline in Mini-Mental State Exam (MMSE) at 12 Months | Assessed for endpoint at Screening/Baseline and 12-Month clinic visits
  Cognition as measured by MMSE (total score possible from 0-30, where a lower score is more affected by Alzheimer's disease)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Kern, Principal Investigator — Cognito Therapeutics
Locations (53):
- United States (53):
  - Barrow Neurological Institute, Phoenix, Arizona
  - CCT Research - Foothills Research Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Advanced Research Center, Inc, Anaheim, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neurology Center of North Orange County, Fullerton, California
  - Syrentis Clinical Research, Santa Ana, California
  - Office of Elizabeth Zarate-Rowell, MD, Seal Beach, California
  - Mile High Research Center, Denver, Colorado
  - JEM Research Institute, Atlantis, Florida
  - South Lake Pain Institute, Clermont, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Charter Research - Lady Lake, Lady Lake, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Coastal Family Medicine - Orange Park, Orange Park, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group - Sarasota, Sarasota, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Brain Matters Research (Kane Center), Stuart, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research - Winter Park, Winter Park, Florida
  - Emory Alzheimer's Disease Research Center, Atlanta, Georgia
  - NeuroStudies, Decatur, Georgia
  - Great Lakes Clinical Trials- Flourish Research- Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials- Flourish Research- Gurnee, Gurnee, Illinois
  - Northern Light Acadia Hospital, Bangor, Maine
  - Boston Center for Memory, Newton, Massachusetts
  - Office of Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Sisu BHR, LLC, Springfield, Massachusetts
  - QUEST Research Institute, Farmington, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - Alzheimer's Memory Center - AMC Research, Matthews, North Carolina
  - Insight Clinical Trials, LLC, Beachwood, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Prisma Health Neurology, Columbia, South Carolina
  - Coastal Neurology, Port Royal, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - North Texas Clinical Trials, Fort Worth, Texas
  - UT Health San Antonio, Glenn Biggs Institute for Alzheimer's and Neurodegenerative Diseases, San Antonio, Texas
  - TRS Health, Stafford, Texas
  - Mercury Clinical Research, Sugar Land, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - ReCogniton Health, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No